CLINICAL TRIAL: NCT00825578
Title: Comparative Study of Bronchoscopic Lung Volume Reduction to Evaluate Relative Efficacy in Patients With Non-Upper Lobe Emphysema
Brief Title: Use of Endobronchial Valves in Non-Upper Lobe Heterogeneous Emphysema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08/H0708/84
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Heterogeneous Emphysema
Keywords: intrabronchial valve; heterogeneous emphysema; non-upper lobe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Upper-lobe predominant emphysema
  Interventions: Device: Intra-bronchial valve (Spiration IBV)
- 2 (Active Comparator): Non-upper lobe predominant emphysema
  Interventions: Device: Intra-bronchial valve (Spiration IBV)

INTERVENTIONS:
Device: Intra-bronchial valve (Spiration IBV) — Device: Intra-bronchial valve (Spiration IBV) The IBV is comprised of a Nitnol frame and a polymer membrane, which is held against the airway mucosa by six elastic struts and will expand and contract with airway movement during breathing. The valve is designed to conform to the size and shape of the airways. The frame has 5 flexible anchors that gently secure to the mucosal wall at a controlled depth. Valves are available in 5, 6 and 7mm diameters appropriate for different airways. During a minimally invasive procedure, a catheter is passed through a bronchoscope (a flexible tube passed into the airways through the mouth) to deploy the umbrella-shaped valves into the airways. Only flexible bronchoscopy equipment is required. The valves are designed to be removed if indicated.
  Other Names: Spiration IBV

SUMMARY:
Hypothesis: Patients with advanced emphysema with predominance of the disease in areas other than the upper lobes, as determined by high resolution computed tomography (HRCT), could have a positive response to valve treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Ex-smoker with smoking cessation confirmed by exhaled carbon monoxide (CO) levels
* Moderate to severe airflow obstruction FEV1 <50% Predicted
* Severe dyspnoea - mMRC ≥2
* Hyperinflation - total lung capacity (TLC) ≥100% predicted, RV ≥150% predicted
* SWT ≥75m
* Optimum COPD treatment for at least 6 weeks
* No COPD exacerbation for at least 6 weeks
* Less than 4 admissions for exacerbation in the preceding 12 months

Exclusion Criteria:

* Patient unable to provide informed consent
* Patient without clear targets for airflow re-distribution
* Total lung CO uptake (TLCO) <15% predicted and FEV1 <15% predicted
* pO2 on air <6.0kPa
* pCO2 on air >8.0kPa
* Neurological, rheumatological or other cause of exercise limitation
* Other major medical illness, e.g. lung cancer that will limit participation
* Production of purulent sputum more often than not (more than 50% of days)
* Clinically significant bronchiectasis
* Large bulla - more than 1/3 of hemithorax volume (i.e. where bullectomy would be more suitable) on CT scan
* Arrhythmia or cardiovascular disease that poses a risk during procedure or exercise
* Prednisolone dose greater than 15mg a day
* Significant pulmonary hypertension - RVSP ≥45mmHg
* Left ventricular failure - left ventricular ejection fraction <45% or left ventricular fraction shortening <23%
* Prior LVRS or lobectomy
* Lung nodule requiring surgery
* Subject completed or is participating in a standard pulmonary rehabilitation program within 3 months of enrolment
* Female of childbearing age with positive pregnancy test
* Subject participated in a research study of investigational drug or device in prior 30 days
* Subject taking clopidogrel, warfarin, or other anticoagulants and unable to abstain for 5 days pre-procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To estimate the difference between study arms in volume changes of the treated lobe(s) by CT scan | 6 months

SECONDARY OUTCOMES:
To estimate the difference between study arms in volume changes of the non-treated lobes by CT scan | 6 months
To estimate the difference between study arms in residual volume | 6 months
To estimate the difference between study arms in FEV1 | 6 months
To estimate the difference between study arms in gas transfer | 6 months
To estimate the difference between study arms in modified MRC dyspnoea score | 6 months
To estimate the difference between study arms on a 6 minute walk test | 6 months
To estimate the difference between study arms in disease specific health status | 6 months
To estimate the difference between study arms in dynamic hyperinflation during cycle ergometry | 6 months
To estimate the difference between study arms in changes in respiratory and quadriceps muscle strength | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pallav Shah, MBBS, MD, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton Hospital, London, United Kingdom